CLINICAL TRIAL: NCT01395160
Title: Female Experiences and Brain Activity: an EEG Investigation Across Psychiatric Disorders
Brief Title: Female Experiences and Brain Activity
Acronym: FEBA
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Glenn Mould, Project Coordinator, King's College London
Other Study IDs: 11/LO/0438
Record Dates: First submitted 2011-05-20; First posted 2011-07-15 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Attention Deficit Hyperactivity Disorder; ADHD; Bipolar Disorder
Keywords: Attention deficit hyperactivity disorder; ADHD; Bipolar Disorder; Electrophysiological; EEG; ERP; Attention; Motivation; Mood instability
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buccal swab samples will be collected for DNA extraction.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adult ADHD
- Bipolar Disorder
- Healthy control

SUMMARY:
The Female Experiences and Brain Activity study will investigate how different groups of people process information in different ways. Using electro-physiological methods it will investigate differences in brain activity between women with ADHD, women with bipolar disorder and those without a psychiatric illness. It will also investigate the relationship between patterns of brain activity, mood and functioning.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) and bipolar disorder (BD) affect approximately 2.5% and 1%, respectively, of the adult population in the UK. They represent a major clinical and economic burden on society. Genetic and environmental risk factors (such as life events for BD); have been identified for each disorder. Despite the highly different symptom presentations for ADHD and BD, it has recently become clear that they share a cognitive characteristic, observed in high response time variability (RTV). This has led to the question of whether the increased RTV, which reflects short-term fluctuations in performance, is a non-specific marker for psychopathology or whether the causes for the higher RTV could differ across disorders. RTV has been identified as a possible early marker of psychopathology; therefore a better understanding of the underlying mechanisms could lead to improved diagnosis and prevention of negative consequences. Further, it will give insight into the comorbidity observed between ADHD and BD. This study will use cognitive-electrophysiological methods to investigate the causes for RTV and its association with other cognitive and neurophysiological impairments observed in each disorder (aim 1). The second question will address whether, within each disorder, current cognitive functioning relates to the patients' current social functioning (aim 2). Adverse life events and other psychosocial risk factors can contribute to high variability in the level of social functioning observed, within and between individuals, in each disorder; yet our understanding of the association between current social functioning and cognitive functioning is limited. Finally the study will explore if any cognitive differences detected by electrophysiological investigation are associated with any candidate gene markers for either disorder (aim 3).

ELIGIBILITY:
Inclusion Criteria:

* current clinical diagnosis of adult ADHD
* or current clinical diagnosis of Bipolar Disorder
* or no history of psychiatric illness
* white European descent

Exclusion Criteria:

* presence of a neurodevelopmental disorder
* epilepsy
* brain injury
* dyslexia
* limited proficiency in English language
* IQ<70
* any current psychiatric medication use (with the exception of mood stabilisers or stimulant medication in the clinical groups)

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population will be recruited through primary care clinics and existing research participant databases.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
cognitive-electrophysiological recordings | 2 hours
  Amplitude and latency of ERP components recorded by 64 scalp electrodes will be compared across groups. Comparison will be carried out by different types of ERP eliciting stimuli (target, non-target, novel, cue etc) from four different paradigms (ERN, CPT-OX with flankers, Fast-task, Novelty Oddball).
Emotional and functional difficulties trait scores | 2 weeks
  Measures assessing ADHD/biploar symptoms traits, mood lability, and functional impairment will be used to generate an index of emotional regulation difficulties and resulting functional impairments. These will be be compared across groups and correlated with the primary ERP outcome measure.

SECONDARY OUTCOMES:
Genotype data from buccal swab samples | 4 hours
  Extracted DNA will be genotyped for genetic markers (SNPs). Depending on results of the primary outcome measures, this information could be used to identify genetic regions associated with observed ERP deficits.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Asherson, MRCPsych, PhD, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - South London and Maudsley NHS Trust, London, London
  - Institute of Psychiatry, King's College London, London, London